CLINICAL TRIAL: NCT03102840
Title: Cross-sectional Study to Establish the Point Prevalence of Serotype 19A Pneumococcal Nasopharyngeal Carriage of Fully Vaccinated Children Aged 6-48 Months 7 Years Following Introduction of PCV-13
Brief Title: Understanding Pneumococcal Carriage and Disease 2017-2020
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: OVG 2017/03
Record Dates: First submitted 2017-03-30; First posted 2017-04-06 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Streptococcus Pneumoniae Infection; Streptococcus Pneumoniae, Invasive Disease; Streptococcal Pneumonia
Keywords: Carriage; Immunogenicity; Pneumococcal conjugate vaccine 13 (PCV 13); Children; Pneumococcus
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bacteria grown from nasopharyngeal swabs Serum to measure serotype specific antibodies levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children nasal swab only: Pneumococcal nasopharyngeal carriage in children aged 6-48 months who have previously received PCV13
  Interventions: Diagnostic Test: Nasopharyngeal swab
- Children nasal swab + serum: Pneumococcal nasopharyngeal carriage and immunogenicity in children aged 6-48 months who have previously received PCV13
  Interventions: Diagnostic Test: Nasopharyngeal swab; Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab — Nasopharyngeal swab will be performed in all participants
Diagnostic Test: blood sampling — Blood sampling will be done by finger-prick in a sub-set of participants
  Groups: Children nasal swab + serum

SUMMARY:
Streptococcus pneumoniae is a type of bacteria that is carried (lives) in the nose of most individuals and can sometimes go on to cause severe infections such as meningitis and pneumonia. There are over 100 types of pneumococcus, and children in the UK have been routinely immunized against pneumococcal disease since 2006. A vaccine against 13 types of pneumococcus (PCV 13) was introduced into the UK in 2010, replacing a previous version that prevented 7 types.

Pneumococcal carriage in the Thames Valley region has been studied over the last 7 years with carriage rates having been shown to be reflective of potential severe pneumococcal disease and hence vaccine effect.

The main purpose of this study is to see whether the pneumococcal immunization program has changed the frequency and nature of pneumococcal bacteria carried by children, as this may give a clue as to what changes in pneumococcal disease are likely to be seen in the future. In addition, this study is especially timely given the possibility of a change in the PCV 13 immunization schedule that is currently being assessed in the 'Sched3' Immunization study (NCT02482636). Obtaining accurate baseline data will be important in informing the interpretation of any subsequent data on carriage rates obtained following introduction of the new schedule.

This study will enrol up to 1600 children aged 13 to 48 months living in the Thames Valley and South Midlands and which have had three doses of 13-valent pneumococcal conjugate vaccine. In addition, up to 800, 6-12 month old children who have received a priming dose of PCV13 will be recruited. The study consists of one visit done at a convenient venue (GP surgeries, educational/ play settings, or home) where a single nasal swab and an optional finger-prick blood sample for a sub-set of 632 participants, will be performed. No additional follow-up is needed. The study recruitment period will be from 2017 onwards.

DETAILED DESCRIPTION:
This is a cross sectional observational study to determine the point prevalence of pneumococcal carriage in children. In this study up to 1600, healthy children aged 13-48 months who have received a complete course of PCV13 at least one month prior to study enrolment, will be recruited. In addition, up to 800, 6-12 month old children who have received a priming dose of PCV13 will be recruited.

For the 13-48 month cohort, an interim analysis for futility to demonstrate an increase in serotype 19A will be performed after the first 750 participants.

The study will be carried out in the Thames Valley and South Midlands. Parents/legal guardians will be approached either by website based advertisements, social media, poster advertisements and emailing and/or handing out information booklets through their child's nurseries, GP Surgeries and educational/play settings. The investigators may also identify potential participants by mailing out invitation letters and leaflets to age appropriate children via the Open Exeter system of National Health Application and Infrastructure Services, the Child Health Computer Department, equivalent NHS database or through the Clinical Research Network. Parents/legal guardians of potential participants who have expressed interest will be directed to the Oxford Vaccine group (OVG) website where they will be able to access the participant information booklet and if appropriate complete online self-screening. If parents approach OVG to express interest, the information booklet will be sent to them and they may be telephone screened.

This study will involve a one off visit. The study visit will be arranged to occur in a convenient venues such as: hospital out patients, university clinic rooms, village halls, church halls, nurseries, participant's homes, sporting and recreational areas, GP practices and other similar venues where pre-school children frequently attend. Permission would be seek from the above venues to carry out any study procedures on their premises. Pre-arranged dates and times will be offered to parents/legal guardians by online booking, phone call or email.

During the visit the investigators would go through the details of the study and provide an opportunity for further questions. For those willing to proceed the investigators would then ask participants to sign a consent form and collect demographic information. A nasopharyngeal swab will be taken, and if consented to do so an optional blood sample will be performed in a subset of 632 participants. No further visits or follow-up will be required.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/guardian of participant is willing and able to give informed consent for participation in the study.
2. In good health as determined by a brief medical history and/or clinical judgement of the investigator.
3. For children aged 13-48months, they must have received three doses of PCV13 as per infant immunization schedule (as confirmed by red book or through vaccination history and age). For children aged 6-12months, they must have received 2 doses of PCV12 as per the infant immunisation schedule.

   (Vaccination history is confirmed by the child's GP or CHCD. The visit and sampling may still proceed if the vaccination history has not been confirmed beforehand and the participant can be subsequently excluded if they were found to not have received all required doses of PCV13.)
4. Aged 13-48 months and at least 28 days since their third PCV13 vaccination or aged 6-12months and at least 28days since their second dose of PCV13.
5. Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

1. Parent/legal guardian unwilling or unable to give written informed consent to participate in the study.
2. Parent/legal guardian less than 18 years of age at time of enrolment.
3. Parent/legal guardian is listed on the study delegation log.
4. Children who were known to be un-immunized or have an incomplete course of PCV13.
5. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
6. History of bleeding disorder.

Temporary exclusion criteria:

1. Febrile illness or temperature of 38°C or above on the day of the visit or in the preceding 24 hours.
2. Respiratory illness on the day of the study visit or in the preceding 24 hours. A respiratory illness will be classified as a combination of at least two of the following symptoms: cough, sore throat, and runny nose.
3. Administration of antibiotics in the month prior to sampling.
4. History of an acute nose bleed (within the last 24 hours), or recent (within the last 3 months) nasal/craniofacial surgery.
5. Receipt of blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 90 days.

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1600 children aged 13 to 48 months, who have received 3 doses of PCV13 800 children aged 6-12 months, who have recieved 2 doses of PCV13
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Serotype 19A-specific carriage rate in healthy children aged 6 to 48 months in 2017-2020. | 3 year
  To determine the serotype 19A-specific carriage rate in healthy children aged 6 to 48 months in 2017-2020, seven years following introduction of PCV13 and to compare this to carriage rates observed in 2014/2015 (OVG 2013/05 study).

SECONDARY OUTCOMES:
To determine the PCV13 vaccine-type pneumococcal serotype-specific nasopharyngeal (NP) carriage rate and serotype distribution in children aged 13 to 48 months who have received a full course of PCV13 | 3 year
  Presence of PCV13 vaccine type pneumococcal serotypes NP swab samples by microarray analysis
To determine the non-PCV vaccine type pneumococcal serotype-specific NP carriage rate and serotype distribution in children aged 6 to 12 months who have received a primary course of PCV13 | 3 years
  Presence of PCV13 non-vaccine type pneumococcal serotypes on NP swab samples by microarray analysis
To determine PCV-13 serotype specific anti-pneumococcus antibody concentrations in fully immunised 6 to 48 month old children | 3 years
  Antibody concentration by ELISA (finger-prick blood sample) for PCV13 vaccine-types

OTHER OUTCOMES:
To compare PCV-13 serotype specific anti-pneumococcal antibody concentrations in age matched, fully immunized 6 to 48 month old children to historical cohorts from the OVG 2013/05 study. | 3 years
  Antibody concentration by ELISA (finger-prick blood sample) for PCV13 vaccine-types obtained in current study and biobank samples of historical cohorts
To assess for carriage of multiple pneumococcal strains in participants in the current study and on stored samples from OVG 2013/05 study. | 3 years
  Microarray analysis of culture 'sweeps' obtained in the current and OVG 2013/05 studies

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiley KS, Ratcliffe H, Voysey M, Jefferies K, Sinclair G, Carr M, Colin-Jones R, Smith D, Bowman J, Hart T, Kandasamy R, Hinds J, Gould K, Berbers G, Tcherniaeva I, Robinson H, Plested E, Aley P, Snape MD. Nasopharyngeal Carriage of Pneumococcus in Children in England up to 10 Years After 13-Valent Pneumococcal Conjugate Vaccine Introduction: Persistence of Serotypes 3 and 19A and Emergence of 7C. J Infect Dis. 2023 Mar 1;227(5):610-621. doi: 10.1093/infdis/jiac376. PMID 36130327